CLINICAL TRIAL: NCT04231123
Title: Pericapsular Nerve Group Block for Analgesia After Hip Arthroplasty: a Randomized Double-Blind, Placebo-Controlled Trial.
Brief Title: Pericapsular Nerve Group Block for Elective Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Tivoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2019/482; 2019-001956-21 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
Keywords: Elective Hip Surgery; PENG Block
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Injected solutions will be prepared by an anesthetist not involved in the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): PENG block with 20 ml of a mixture of 1% Lidocaine with 0,5% Ropivacaine and 1/400.000 Epinephrine
  Interventions: Procedure: PENG Block with local anesthetic
- Placebo group (Placebo Comparator): PENG block with 20 ml of 0,9% saline
  Interventions: Procedure: PENG Block with 0,9% saline

INTERVENTIONS:
Procedure: PENG Block with local anesthetic — After induction of general anesthesia, PENG block with 20 ml of a mixture of 1% Lidocaine with 0,5% Ropivacaine and 1/400.000 Epinephrine will be performed as described by Giron-Arongo et al with a high frequency linear probe. A 22G 80 mm needle (SonoPlex, Pajunk ) will be used.
  Arms: PENG group
Procedure: PENG Block with 0,9% saline — After induction of general anesthesia, PENG block with 20 ml of 0,9% saline will be performed as described by Giron-Arongo et al with a high frequency linear probe. A 22G 80 mm needle (SonoPlex, Pajunk ) will be used.
  Arms: Placebo group

SUMMARY:
This study examine the effect of Pericapsular Nerve Group (PENG) Block on analgesia after elective hip arthroplasty. Half of participants will receive a PENG Block with local anesthetic, while the other half will receive a PENG Block with a placebo.

DETAILED DESCRIPTION:
Optimized analgesia is crucial for early mobilization after hip arthroplasty. Regional anesthesia, like fascia iliaca block or femoral nerve block, have limited indication because of motor blockade whereas local infiltrations analgesia have shown conflicting analgesic efficacy results in hip arthroplasty.

Pericapsular nerve group (PENG) block is a new regional anesthesia technique targeting specifically sensory nerve branches of the hip articulation. It has been originally described in hip fracture patients.

The aim of this study is to evaluate the efficacy of PENG block on analgesia after elective hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty
* General anesthesia
* Enhanced Recovery Program

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Score > 2
* Drug allergy
* Significant psychiatric disturbances
* Preoperative opioid use
* Contraindication to acetaminophen, celecoxib, methylprednisolone or tranexamic acid
* Body Mass Index > 40 kg/m²

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain Score on first Mobilization | Postoperative time until midnight day 0
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on first mobilization at day 0 after surgery

SECONDARY OUTCOMES:
Maximum Pain Score in Post-Anaesthesia Care Unit | Through postoperative time during Post Anesthesia Care Unit stay at day 0
  Maximum Pain score evaluated in Post Anesthesia Care Unit by a a visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
Morphine Consumption at Day 0 | Postoperative time until midnight day 0
  Total of Piritramid, Oxycodone and Oxycodone Extended Released expressed as equivalent of morphine at day 0
Piritramid Consumption | Through the end of surgery until Post Anesthesia Care Unit discharge to the ward at day 0
  Total of Piritramid use from the end of surgery until Post Anesthesia Care Unit discharge to the ward
Morphine Consumption at Day 1 | Postoperative time during Post Anesthesia Care Unit stay at day 0
  Total of Oxycodone and Oxycodone Extended Released expressed as equivalent of morphine at day 1
Morphine Consumption at Day 2 | Postoperative time until midnight day 2
  Total of Oxycodone and Oxycodone Extended Released expressed as equivalent of morphine at day 2
Pain Score at Rest 2h Postop | 2 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest 2h after surgery
Pain Score on mobilization 2h Postop | 2 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization 2h after surgery
Pain Score at Rest 4h Postop | 4 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest 4h after surgery
Pain Score on mobilization 4h Postop | 4 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization 4h after surgery
Pain Score at Rest 6h Postop | 6 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest 6h after surgery
Pain Score on mobilization 6h Postop | 6 hours after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization 6h after surgery
Pain Score at Rest Day 1 AM | Day 1 in the morning after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest in the morning of day 1
Pain Score on mobilization Day 1 AM | Day 1 in the morning after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization in the morning of day 1
Pain Score at Rest Day 1 PM | Day 1 in the afternoon after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest in the afternoon of day 1
Pain Score on mobilization Day 1 PM | Day 1 in the afternoon after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization in the afternoon of day 1
Pain Score at Rest Day 2 AM | Day 2 in the morning after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest in the morning of day 2
Pain Score on mobilization Day 2 AM | Day 2 in the morning after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization in the morning of day 2
Pain Score at Rest Day 2 PM | Day 2 in the afternoon after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain at rest in the afternoon of day 2
Pain Score on mobilization Day 2 PM | Day 2 in the afternoon after surgery
  A visual analog pain scale anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) will be used to evaluate pain on mobilization in the afternoon of day 2
First Mobilization Success | Postoperative time until midnight day 0
  Success rate of patients mobilized the day of surgery
Mean remifentanil Infusion Rate | Intraoperatively
  Total infused remifentanil dose per kg body weight per minute of total operative time
Quadriceps weakness | Through postoperative time during Post Anesthesia Care Unit stay at day 0
  Evaluation of quadriceps motricity by Neal test which consist in supporting the knee under the popliteal fossa and asking the patient to extend the knee against resistance.

OTHER OUTCOMES:
Patient satisfaction after 24h | 24 hours after surgery
  Patient satisfaction for the first 24h after surgery recorded with a scale from 0 (unsatisfied) to 10 (extremely satisfied).
Length of hospital stay | During hospital stay, up to 1 week
  Calculated as the number of days between the hospital admission and discharge dates.
PACU stay | Postoperative time during Post Anesthesia Care Unit stay at day 0
  Time from the arrival in Post Anesthesia Care Unit until discharge to the ward
Postoperative Nausea and Vomiting | PACU, at 2, 6, 24, and 48 hours
  The incidence and severity of postoperative nausea (none=0, mild=1, moderate=2, severe=3), episodes of vomiting, and need for rescue antiemetics was also documented.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Van Rompaey, MD, Principal Investigator — Centre Hospitalier Universitaire de Tivoli
Locations (1):
- Chu Tivoli, La Louvière, Belgium

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657